CLINICAL TRIAL: NCT07307794
Title: Characterisation of Adhesion Performance of a Newly Developed Esflurbiprofen Topical System (EFTS) - a Phase I, Open-label Study in Healthy Subjects.
Brief Title: To Evaluate the Adhesion of TK-254RX on Healthy Participants
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Teikoku Seiyaku Co., Ltd. (Industry)
Collaborators: SocraTec R&D GmbH (Other); SocraMetrics GmbH (Industry); HWI pharma services GmbH (Industry); Clinsearch GmbH (Unknown); CRM Biometrics GmbH (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TK-254RX-0107; 2025-523577-42-00 (EU CTIS Number)
Record Dates: First submitted 2025-12-15; First posted 2025-12-29 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Healthy Participants

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- TK-254RX (Experimental): TK-254RX will be applied to the left or right lower leg above the ankle once daily over 3 consecutive days
  Interventions: Drug: Esflurbiprofen Topical System

INTERVENTIONS:
Drug: Esflurbiprofen Topical System — The total of one TK-254RX per day for 3 days

SUMMARY:
This study is a single-center, open-label, multiple-dose trial in healthy participants. The primary purpose of this study is to assess the adhesion of TK-254RX. Secondary purposes are to assess the safety of TK-254RX and the residual amount of the patch.

ELIGIBILITY:
Inclusion Criteria:

* age: 18 to 64 years
* good state of health
* written informed consent, after having been informed about benefits and potential risks of the clinical trial, as well as details of the insurance taken out to cover the participants enrolled in the clinical trial

Exclusion Criteria:

* any injury of body which may induce the restriction of body movement
* excessively hairy skin at application site
* current or anamnestic known skin disorder (e.g., atopic dermatitis (eczema), neurodermatitis, contact allergy, psoriasis, vitiligo, melanoma, squamous cell carcinoma) or shaving hair at application site, which might interfere with the safety or tolerability of the active ingredient
* history of excessive sweating/hyperhidrosis inclusive of application site
* participation in a clinical study within 30 days before inclusion in the study or concomitantly
* drug or alcohol abuse in the opinion of the investigator
* pregnant and lactating women
* women of child-bearing potential (WOCBP) who do not agree to apply highly effective contraceptive methods

  * Surgical sterilization
  * Hormonal contraception: combined (estrogen and progestogen containing) hormonal contraception, e.g., oral, intravaginal, transdermal, and progestogen-only hormonal contraception e.g. oral, injectable, implantable as well as intrauterine device (IUD) and intrauterine hormone-releasing system (IUS) each in combination with male condom to increase safety effect (double barrier method))
  * Bilateral tubal occlusion
  * Total abstinence throughout the study at the discretion of the Investigator
  * Periodic abstinence is not an acceptable method of contraception. An acceptable method of contraception must be maintained throughout the study.
  * A woman who is post-menopausal and not surgically sterile must have a negative urine pregnancy test at screening but will not need to comply with an acceptable method of contraception. Women are considered post-menopausal and not of childbearing potential if they had 12 months of natural (spontaneous) amenorrhea with an appropriate clinical profile (e.g., age appropriate, history of vasomotor symptoms) or six months of spontaneous amenorrhea with serum FSH levels > 40 mIU/mL or had surgical bilateral oophorectomy (with or without hysterectomy) at least six weeks ago. In the case of oophorectomy alone, only when the reproductive status of the woman had been confirmed by follow up hormone level assessment.
* known hypersensitivity to Esflurbiprofen, R-flurbiprofen or one of the excipients of the EFTS
* existing cardiac and/or hematological diseases or pathological findings, which might interfere with the safety or tolerability of the active ingredient
* existing hepatic and/or renal diseases or pathological findings, which might interfere with the safety or tolerability of the active ingredient
* known liver or kidney insufficiency
* existing gastrointestinal diseases or pathological findings, which might interfere with the safety or tolerability of the active ingredient
* history of relevant CNS and/or psychiatric disorders and/or currently treated CNS and/or psychiatric disorders
* systolic blood pressure < 90 or > 139 mmHg
* diastolic blood pressure < 60 or > 89 mmHg
* pulse rate < 50 bpm or > 90 bpm
* ECG assessment by investigator: "conspicuous"
* participants who use any impermissible treatment or for whom restrictions apply
* subject is vulnerable such as detained or committed to an institution by a court of law or by legal authorities or close affiliation with the sponsor or the investigational site (e.g., a close relative of the investigator, dependent person (e.g., employee of or student at the investigational site), employee of the sponsor or affiliates)
* subjects who have experienced asthma, urticaria, or allergic-type reactions after taking aspirin or other NSAIDs
* subject with known bronchial asthma from previous history
* Laboratory values are out of normal range

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 90 (Estimated)
Dates: Start 2026-01-19 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Characterization of the patch adhesion | Day 1 to Day 4
  Measuring the patch adhesion area by percentage visually by site staff, with the patch remaining adhered

SECONDARY OUTCOMES:
Recording adverse events and serious adverse events | Day 1 to Day 4
  Characterization of the occurrence of adverse events or serious adverse events of TK-254RX
Residual amount of S-flurbiprofen | Day 3 to Day 4
  Residual amount of S-flurbiprofen in the used patch applied on Day 3

CONTACTS AND LOCATIONS:
Overall Officials: Kenichi Nishiyama, Study Chair — Teikoku Seiyaku Co., Ltd.
Locations (1):
- Deutsche Sporthochschule Köln, Am Sportpark Muengersdorf 6, Clogne, Germany

IPD SHARING:
Plan to Share IPD: No